CLINICAL TRIAL: NCT04376814
Title: The Regimen of Favipiravir Plus Hydroxychloroquine Can Accelerate Recovery of the COVID-19 Patients With Moderate Severity in Comparison to Lopinavir/Ritonavir Plus Hydroxychloroquine Regimen: an Open-label, Non-randomized Clinical Trial Study
Brief Title: Favipiravir Plus Hydroxychloroquine and Lopinavir/Ritonavir Plus Hydroxychloroquine in COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Responsible Party: Principal Investigator, Mohammad Sadegh Bagheri Baghdasht, Principal Investigator, Baqiyatallah Medical Sciences University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR.BMSU.REC.1399.017
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Favipiravir; Kaletra; Hydroxychloroquine; Lopinavir/Ritonavir
MeSH Terms: conditions — COVID-19 | interventions — favipiravir; Hydroxychloroquine; Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): In this group, Patients will be given a stat dose of 1600mg Favipiravir tablets for the first time, and for next time they will be given 600mg of favipiravir tablets three times per day for 7 days, plus 200mg of Hydroxychloroquine two times per day will be given to patients for 7 days.
  Interventions: Drug: Favipiravir; Drug: Hydroxychloroquine
- Control Group (Active Comparator): In this group, Patients will be given a stat dose of 400mg Hydroxychloroquine tablets plus 200/50 mg of Lopinavir/Ritonavirtwo times per day for seven days.
  Interventions: Drug: Hydroxychloroquine; Drug: Lopinavir / Ritonavir

INTERVENTIONS:
Drug: Favipiravir — Patients will be given a stat dose of 1600mg Favipiravir tablets for the first time, and for next time they will be given 600mg of favipiravir tablets three times per day for 7 days
  Arms: Test Group
Drug: Hydroxychloroquine — 200mg of Hydroxychloroquine two times per day will be given to patients for seven days in Test group, and Patients in Control group will be given a stat dose of 400mg Hydroxychloroquine tablets two times per day.
Drug: Lopinavir / Ritonavir — Patients will be given 200/50 mg of Lopinavir / Ritonavir two times per day for seven days.
  Other Names: Kaletra
  Arms: Control Group

SUMMARY:
This is an open-label, non-randomized clinical trial study. The number of 40 COVID-19 patients with moderate severity will be admitted in progressive care units (PCUs) and intensive care units (ICUs) enrolled in the study. The sampling will be purposive and based on the same independent variables, including age, gender, past medical histories, and the situation of the patient at the admission day, and ventilator support. The patients will be allocated into two groups with different regimens. Group "A" (regimen A)will be defined as Favipiravir 1600 mg a first dose and 600 mg in 3 divided doses daily plus 400 mg in 2 divided doses of Hydroxychloroquine every day. The group "B" (regimen B) will be contained 400 mg of Lopinavir/Ritonavirin 2 divided doses plus the first dose (400 mg) of Hydroxychloroquine. Hydroxychloroquine will not be used for adverse drug reactions. The regimen remained at least 7 up to 10 days.

Data will be analyzed using statistical package for social sciences (SPSS) version 18 (SPSS Inc. Chicago, IL, USA) for windows. The variables will be compared using independent and paired T-test for normally distributed variables and Wilcoxon, Chi-square for non-normal distributed variables. The Kaplan Meier test will be used for survival analysis and the one-sample Kolmogorov-Smirnov test for the evaluation of distributions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 based on either ground glass appearance in chest CT scan or positive RT-PCR test for COVID-19
* Requiring hospitalization
* Patient's age between 16 and 100 years
* Signed informed consent form

Exclusion Criteria:

* Receiving other antiviral medications such as (Kaletra, Ribavirin, Oseltamivir)
* Chronic liver or renal failure
* HIV; GI bleeding
* Pregnancy
* Lactation
* QT interval > 500 ms.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-29 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Mortality | Up to 28 days
  In-hospital mortality
long of hospitalization | Up to 28 days
  long of hospitalization
Laboratory Treatment Response (Blood cell count) | Up to 28 days
  Laboratory Treatment Response; return of blood cell count to normal
Laboratory Treatment Response (CRP ) | Up to 28 days
  Laboratory Treatment Response; return of CRP values to normal
Dyspnea | Up to 28 days
  shortness of breath based on symptoms of Dyspnea and questioning the patient
Oxygen saturation without supplemental oxygen. | Up to 28 days
  Oxygen saturation without supplemental oxygen. Measurement will be done after discontinuation of oxygen therapy for 5 minutes.
Oxygen therapy | Up to 28 days
  Oxygen therapy maximum flow during the day (lit/min)

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Sadegh Bagheri Baghdasht, Tehran, Iran